CLINICAL TRIAL: NCT00656877
Title: Incidence of Fat Embolism With Computer Assisted Total Knee Arthroplasty
Acronym: Fat Embolism
Status: Completed | Type: Observational
Sponsor: Marshall University (Other)
Responsible Party: Ali Oliashirazi, MD, Marshall University School of Medicine
Other Study IDs: 6077
Record Dates: First submitted 2007-12-27; First posted 2008-04-11 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Fat Embolism Syndrome
Keywords: Fat Embolism Total Knee Arthroplasty
MeSH Terms: conditions — Embolism, Fat

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
The study to determine the if the incidence of Fat Embolism is decreased using Computer Assisted technology when performing a Total Knee Arthroplasty.

DETAILED DESCRIPTION:
Computer assisted total knee arthroplasty is at its inception currently. There are many unknowns about this specific technique, particularly when it comes down to fat embolism syndrome. There is a high incidence of fat embolism during total knee arthroplasty as seen both by echocariography as well as sampling of right atrial blood. During a jig-based, or traditional, total knee arthroplasty, a rod is placed inside the femur, and sometimes the tibia as well. Intrusumentations of the medullary canal is known to cause fat embolism. Fat embolism is a syndrome which can produce post-operative confusion, hypoxemia, all the way to post-op and intra-operative death.

Computer assisted total knee arthroplasty does not use intramedullary jigs. It is presumed that by not instrumenting the medullary canal, the rate of fat embolism will be significantly reduced.

Fifty patient s will be studied while they are having a computer assisted total knee arthoplasty. A PICC line will be placed in their arm by an interventional radiologist pre-operatively. This PICC line will be thread into the right atrium. Right atrial blood will be sent to pathology every 10 minutes during the 60 to 90 minute procedure and at intervals post-op. The right atrial blood will be stained for bone marrow elements.

This study is to presumed to show yet another benefit of computer assisted surgery.

ELIGIBILITY:
Inclusion Criteria:

* Must be a candidate for Computer Assisted Total Knee Arthroplasty

Exclusion Criteria:

* Mentally incompetent patients excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are deemed candidates for Computer Assisted Total Knee Arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Oliashirazi, MD, Principal Investigator — Marshall University
Locations (1):
- Marshall University School Of Medicine, Department of Orthopaedics, Huntington, West Virginia, United States